CLINICAL TRIAL: NCT02396823
Title: Respiratory Motor Control and Blood Pressure Regulation After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander V Ovechkin, MD, PhD, Associate Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OICB101489; R01HL103750-01A1 (NIH)
Record Dates: First submitted 2015-02-24; First posted 2015-03-24 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
Keywords: Blood pressure regulation; Respiratory Muscle Training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory Muscle Training (Experimental): Each training session will last about 45-60 min and will occur five times weekly during one month. During the RMT sessions, the patient will remain in their personal wheelchair. They will be asked to breath through a special device with regulated resistance to breathing air. In the 20 sessions starting from the lowest resistance, the goal will be to train the muscles they use to breathe by slowly increasing this resistance. They will perform six work sets, 5 minutes in duration, separated by rest intervals lasting 1-3 minutes.
  Interventions: Behavioral: Respiratory Muscle Training
- Control (No Intervention): Following screening process and recruiting, subjects from both Healthy Control and SCI Control groups will undergo the same procedures as subjects from SCI group excluding the training intervention.

INTERVENTIONS:
Behavioral: Respiratory Muscle Training — Standard threshold Positive Expiratory Pressure Device and threshold Inspiratory Muscle Trainer assembled together using a T-shaped connector with flanged mouthpiece will be used. The participants will be instructed to perform inspiratory and expiratory efforts against a resistive load. Training session lasts 45 minutes per day, 5 days per week, for 4 weeks.
  Arms: Respiratory Muscle Training

SUMMARY:
The proposed study is designed to answer a novel research question: Can resistive respiratory muscle training designed to improve respiratory motor control also improve blood pressure regulation impaired by spinal cord injury? Resistive breathing exercise, or respiratory muscle training, has been applied to rehabilitate breathing after spinal cord injury, but has not been evaluated as a method for increasing resting blood pressure and / or improving its regulation under stress as is planned in the proposed project. For the first time, respiratory muscle training intervention will be used as a tool to investigate the physiological relationships between pulmonary and cardiovascular function in individuals with Spinal Cord Injury (SCI). Thus, it will foster a new direction from which to address neglected issues surrounding the cardiovascular complications of spinal cord injury.

DETAILED DESCRIPTION:
Screening:

To aid in determining eligibility, participants will have a respiratory and cardiovascular function tests. The participants will also have an ASIA (American Spinal Injury Association) exam to grade the degree and level of their SCI.

Enrollment:

Following screening process, consenting and recruiting, the experimental recordings:

1. Pulmonary Function Test- This test measures lung volumes, airflow and airway pressure with standard equipment;
2. Respiratory Motor Control Assessment- Pulmonary function test is repeated while participant is sitting in a special hospital bed and lying on their back while the investigators record electrical impulses from their neck, chest, arms, legs, abdomen and back muscles. These impulses record how their muscles are contracting. The investigators also record how their chest and abdomen are moving by placing elastic belts around their chest and abdomen. Blood pressure will be measured using a finger cuff;
3. Orthostatic stress test- Using the same methods as above, the investigators will measure blood pressure, heart rate and chest and abdomen movements while the participant is lying down on their back and when the position is suddenly changed to sitting in the investigators' cardiac chair or to upright vertical position on a Tilt table. The investigators will measure blood samples at several intervals from a small catheter inserted into the vein in the arm.
4. Ultrasound of the heart will be performed before and after the Respiratory Muscle Training (RMT) program.

RMT:

During the training session, subjects will be seated in their personal wheelchair with an approximately 45° head-up tilt with nose clip on. Standard threshold Positive Expiratory Pressure Device or standard threshold Inspiratory Muscle Trainer or combination of both will be used to breathe through with adjustable resistance ranging of 20 to 41 cm of water.

All of these devices are in routine clinical use. These devices will be assembled together using a T-shaped connector with flanged mouthpiece. The participants will be instructed to perform inspiratory and expiratory efforts against a resistive load. During inhalation, the subjects will be instructed to sustain the effort until their lungs feel full. During exhalation, the subjects will be instructed to sustain their effort until their lungs feel empty.

This study will use two test-subject pre-training assessment sessions to provide its internal experimental group control. To match the training period (4 weeks), the pre-training assessment sessions will be performed four weeks apart and the measured parameters will be used to establish the variance in untrained subjects. The pulmonary function tests include the measurement of lung volume, airflow, and static mouth airway pressures using standard clinical methods and equipment while the SCI participant is sitting in their personal wheelchair. The investigators will also record the surface electromyogram (sEMG) activity from the trunk muscles during Maximal Inspiratory Pressure (PImax) and Maximal expiratory pressure (PEmax) measurements in supine position (PImax and PEmax tasks). The investigators will measure a Sympathetic Skin Response (SSR) by recording limb skin resistance during neural stimulations. The investigators will assess beat-to-beat systemic blood pressure, heart rate and cardiac output will be recorded during the orthostatic stress test. In addition, during the orthostatic stress test, the investigators will collect venous blood samples to measure the levels of catecholamines. In addition to the beat-to beat calculated, resting cardiac output will be measured by ultrasonic cardiac echography. After these initial tests, participants will be assigned to RMT. The participants in experimental group will complete the study after 4 weeks of training totaling 20 sessions of 45 minutes per day carried out 5 days per week. The testing battery will be repeated immediately after completing the training and repeatedly during the follow-up period. Ten matched control subjects will undergo the same procedures except training.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. stable medical condition without diseases or autonomic dysreflexia that would contraindicate RMT;
3. no painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore or urinary tract infection that might interfere with RMT;
4. no clinically significant depression, psychiatric disorders or ongoing drug abuse;
5. clear indications that the period of spinal shock is concluded determined by presence of muscle tone, deep tendon reflexes or muscle spasms;
6. no current anti-spasticity medication regimen;
7. non-progressive C3-T5 American Spinal Cord Injury Association Designation of A-D SCI;
8. not ventilator dependent for respiration;
9. sustained SCI at least 6 months prior to entering the study;
10. at least 15%-deficit in pulmonary function outcomes (FVC and FEV1) detected by screening spirometry; and
11. orthostatic hypotension (the decrease 20mm Hg or more in systolic or a reduction 10mm Hg or more in diastolic blood pressure on changing body position from a supine to an upright) detected by screening orthostatic stress test

Exclusion Criteria:

1. a presence of major cardiovascular or pulmonary disease, endocrine disorders, malignancy, marked obesity, deep vein thrombosis, and major gastrointestinal problem such as swallowing or other major medical illness contraindicated for respiratory muscle training or testing.
2. Pregnant women are excluded from this study, as the risk to the fetus is unknown. No pregnancy test or birth control regimen will be required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Changes in Pulmonary Function Test outcomes | At baseline, after 1-month long respiratory training, and during 6 months of follow-up period
  Lung volumes, capacities, air flow, and airway pressure assessed using standard spirometry and maximum airway pressure recordings.

SECONDARY OUTCOMES:
Changes in Respiratory Motor Control Assessment outcomes | At baseline, after 1-month long respiratory training, and during 6 months of follow-up period
  Respiratory multi-muscle activation (amplitude and co-activation) assessed using standard surface electromyography.
Changes in Orthostatic Stress Test outcomes | At baseline, after 1-month long respiratory training, and during 6 months of follow-up period
  Beat-to-beat blood pressure, heart rate, and catecholamines variability assessed during standard orthostatic sit-up stress test.
Changes in cardiac output | At baseline, after 1-month long respiratory training, and during 6 months of follow-up period
  Amount of blood pumping through the heart during one minute assessed using standard heart echography.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ovechkin, MD, PhD, Principal Investigator — avovec02@louisville.edu
Locations (1):
- Frazier Rehabilitation and Neuroscience Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared with scientific collaborators for analysis and interpretation.
Supporting Information: Study Protocol, CSR
Time Frame: Pre-processed data will be available from November 2016 to December 2027.
Access Criteria: Deidentified data sets

REFERENCES:
- [Derived] Legg Ditterline BE, Aslan SC, Randall DC, Harkema SJ, Castillo C, Ovechkin AV. Effects of Respiratory Training on Heart Rate Variability and Baroreflex Sensitivity in Individuals With Chronic Spinal Cord Injury. Arch Phys Med Rehabil. 2018 Mar;99(3):423-432. doi: 10.1016/j.apmr.2017.06.033. Epub 2017 Aug 9. PMID 28802811